CLINICAL TRIAL: NCT04286581
Title: Comparison of Ambu Auragain and I-Gel Supraglottic Airways in Adult Patients at an Ambulatory Surgery Center
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: ANES-2020-28604
Record Dates: First submitted 2020-02-24; First posted 2020-02-27 (Actual); Results first posted 2022-12-19 (Actual); Last update posted 2022-12-19 (Actual); Status verified 2022-11

CONDITIONS: Anesthesia; Surgery

STUDY DESIGN:
Intervention Model Description: Patients who are scheduled for elective ambulatory surgery under general anesthesia will be randomized to one of two groups. Group 1 will receive an I-gel laryngeal mask airway (LMA) and group 2 will receive an Ambu Auragain LMA.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Igel Larnygeal Mask Airway (Experimental): Group 1 will receive the I-Gel Laryngeal Mask Airway for airway maintenance during general anesthesia
  Interventions: Device: I-Gel Laryngeal Mask Airway
- Ambu Auragain Laryngeal mask airway (Active Comparator): Group 2 will receive the Ambu Auragain Laryngeal Mask Airway for airway maintenance during general anesthesia
  Interventions: Device: Ambu Auragain Laryngeal Mask Airway

INTERVENTIONS:
Device: I-Gel Laryngeal Mask Airway — The I-Gel Laryngeal Mask Airway is a medical device that keeps a patient's airway open during anaesthesia or unconsciousness.
  Arms: Igel Larnygeal Mask Airway
Device: Ambu Auragain Laryngeal Mask Airway — The Ambu Auragain Laryngeal Mask Airway is a medical device that keeps a patient's airway open during anaesthesia or unconsciousness.
  Arms: Ambu Auragain Laryngeal mask airway

SUMMARY:
The purpose of this study is to determine if an I-gel laryngeal mask airway (LMA) has a higher oropharyngeal leak pressure compared to an Ambu Auragain in adult patients in an ambulatory surgery center.

DETAILED DESCRIPTION:
Patients who are scheduled for elective ambulatory surgery under general anesthesia will be randomized to one of two groups. Group 1 will receive an I-gel laryngeal mask airway (LMA) and group 2 will receive an Ambu Auragain LMA.

ELIGIBILITY:
Inclusion Criteria:

- undergoing outpatient ambulatory surgery under general anesthesia that is amenable to using a laryngeal mask airway

Exclusion Criteria:

* non-English speaking patients
* patients with abnormal airway anatomy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2021-03-22 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Hutchins, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Igel Larnygeal Mask Airway | Ambu Auragain Laryngeal Mask Airway
Started | 74 | 74
Completed | 70 | 70
Not Completed | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Igel Larnygeal Mask Airway | Ambu Auragain Laryngeal Mask Airway | Total
Number analyzed (Participants) | 70 | 70 | 140
Age, Continuous [Mean (Standard Deviation); unit: years] | 45 (16.9) | 44.6 (19) | 44.8 (17.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 34 | 61
  Male | 43 | 36 | 79
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Oropharyngeal Leak Pressure (OLP)
Description: OLP will be measured immediately after insertion. This will be accomplished by closing the expiratory valve while keeping fresh gas flow at 3 liters/minute until equilibrium is reached. Pressure will be reported in cmH2O.
Time Frame: immediately after placement
Measure: Mean (Standard Deviation); unit: cm H20
Arm/Group | Igel Larnygeal Mask Airway | Ambu Auragain Laryngeal Mask Airway
Number analyzed (Participants) | 70 | 70
cm H20 | 20.9 (6) | 22.6 (5.5)

2. Secondary Outcome: Time to Placement
Description: Time required to place laryngeal mask airway will be measured and reported in seconds.
Time Frame: time from opening mouth to successful placement (4 hours)
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | Igel Larnygeal Mask Airway | Ambu Auragain Laryngeal Mask Airway
Number analyzed (Participants) | 70 | 70
seconds | 8.9 [5.3 to 18] | 30.4 [24.6 to 42.5]

3. Secondary Outcome: Sore Throat
Description: Participants will be asked upon discharge from recovery room (approximately 8 hours post surgery) to rate the soreness of their throat on a numerical rating scale of 0-10 (0 being no soreness and 10 being maximum imaginable soreness). Participants will be asked to rate throat soreness again via phone call approximately 24 hours after surgery.
Time Frame: Pain right before discharge from pacu (8 hours)
Measure: Median (Inter-Quartile Range); unit: numerical rating scale
Arm/Group | Igel Larnygeal Mask Airway | Ambu Auragain Laryngeal Mask Airway
Number analyzed (Participants) | 70 | 70
numerical rating scale | 0 [0 to 1] | 0 [0 to 1]

4. Secondary Outcome: Sore Throat
Description: as for outcome 3
Time Frame: 24 hours post-surgery
Measure: Median (Inter-Quartile Range); unit: numerical rating scale
Arm/Group | Igel Larnygeal Mask Airway | Ambu Auragain Laryngeal Mask Airway
Number analyzed (Participants) | 70 | 70
numerical rating scale | 0 [0 to 1] | 0 [0 to 1]

ADVERSE EVENTS:
Description: Total Number of Participants at Risk for serious and other [non-serious] adverse events and all-cause mortality were not collected or assessed as part of the study
Arm/Group | Igel Larnygeal Mask Airway | Ambu Auragain Laryngeal Mask Airway
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-08): https://cdn.clinicaltrials.gov/large-docs/81/NCT04286581/Prot_SAP_000.pdf